CLINICAL TRIAL: NCT03848936
Title: Evaluation of Functional Status and Mental Functions of Adult Cerebral Palsy Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Bilinç Doğruöz Karatekin, MD, Research Assistant of PMR, Istanbul Medeniyet University
Other Study IDs: Medeniyet CP
Record Dates: First submitted 2019-02-04; First posted 2019-02-21 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Cerebral Palsy
Keywords: adult cerebral palsy; cerebral palsy; functional status; mental function
MeSH Terms: conditions — Cerebral Palsy | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adult cerebral palsy patients: >18 age cerebral palsy diagnosed patients evaluated with a survey.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Survey includes age, gender, cerebral palsy type, education, mental status, working status, living conditions, comorbidities, pain, spasticity, contractures, deformities, mobility status and gross motor function classification system level

SUMMARY:
In adult cerebral palsy patients , a questionnaire study will be conducted to determine the functional level and to determine the effect on quality of life. In this survey, age, gender, demographic information of the patient, as well as additional diseases which can be seen together with cerebral palsy will be questioned.

DETAILED DESCRIPTION:
In adult patients diagnosed with cerebral palsy, a questionnaire study will be conducted to determine the functional level and to determine the effect on quality of life. In this survey, age, gender, demographic information of the patient, as well as additional diseases which can be seen together with cerebral palsy will be questioned. There are studies about the functional status of adults with CP in the literature; However, there is no study conducted on this subject in our country. In this study, it was aimed to evaluate the functional status and mental functions of adults with CP who applied to our hospital.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Diagnosed with cerebral palsy
* Who voluntarily participate the study

Exclusion Criteria:

* <18 years old
* Who does not give permission to participate the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cerebral palsy patients
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-02-20 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Functional status of adult cerebral palsy patients | 1 year
  Evaluated with living status (alone/ with family / with / with spouse / with carer)
Functional status of adult cerebral palsy patients | 1 year
  Evaluated with working status (no, part-time, full-time)
Functional status of adult cerebral palsy patients | 1 year
  Evaluated with comorbidities
Functional status of adult cerebral palsy patients | 1 year
  Evaluated with spasticity (yes or no)
Functional status of adult cerebral palsy patients | 1 year
  Evaluated with deformity and contractures ( no, mild, moderate, severe)
Functional status of adult cerebral palsy patients | 1 year
  Evaluated with pain status (yes or no)
Functional status of adult cerebral palsy patients | 1 year
  Evaluated with mobility status ( 5 degrees )
Mental status of adult cerebral palsy patients | 1 year
  Mental status simply classified as normal/minor/moderate/severe mental retardation.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University Faculty of Medicine, Physical Therapy and Rehabilitation Department, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided